CLINICAL TRIAL: NCT01892267
Title: Comparison Outcomes and Complications of Self-Propelled vs. Standard Percutaneous Endoscopic Gastrojejunostomy (PEG-J); a Randomized Single Blind Clinical Trial
Brief Title: Self-Propelled Versus Standard Percutaneous Endoscopic Gastrojejunostomy(PEG-J); RCT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated prematurely as costs incurred were more than the available funds.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Mouen Khashab, Assistant Professor of Medicine; Director of Therapeutic Endoscopy, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NA_00079056
Record Dates: First submitted 2013-07-01; First posted 2013-07-04 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Feeding Tube
Keywords: PEGJ; PEG-J; Percutaneous Endoscopic Gastrostomy; Feeding tube; Gastroparesis; Acute pancreatitis; Stroke; Respiratory failure; GERD; Balloon; Self-propelled
MeSH Terms: conditions — Gastroparesis; Pancreatitis; Stroke; Respiratory Insufficiency; Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self-propelled PEGJ feeding tube (Experimental): Patients in this arm will receive self-propelled balloon PEGJ tube.
  Interventions: Device: PEG-J placement
- Standard PEGJ feeding tube (Active Comparator): Patients in this arm will receive the standard commercially availabel PEGJ tube.
  Interventions: Device: PEG-J placement

INTERVENTIONS:
Device: PEG-J placement — PEG-J placement

SUMMARY:
Our main hypothesis is that self-propelled Percutaneous Endoscopic Gastrojejunostomy tube (PEG-J) that has a balloon on it's tip is associated with lower J-tube retrograde migration rate, and lower rates of short- and long-term complications when compared to standard PEGJ feeding tubes.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult patients (18-80 years of age) with need for post-pyloric feeding (patients unable to eat due to stroke, intubated patients with respiratory failure, patients with acute pancreatitis, etc).
* Ability to give informed consent.

Exclusion Criteria:

* Unable to give informed consent
* Pregnant or breastfeeding women (all women of child-bearing age will undergo urine pregnancy testing)
* Acute gastrointestinal bleeding
* Coagulopathy defined by prothrombin time < 50% of control; PTT > 50 sec, or INR > 1.5), on chronic anticoagulation, or platelet count <50,000
* Inability to tolerate sedated upper endoscopy due to cardio-pulmonary instability or other contraindication to endoscopy
* Cirrhosis with portal hypertension, varices, and/or ascites
* Allergy to egg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-09-06 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mouen Khashab, MD, Principal Investigator — Johns Hopkins Hospital Department of Gastroenterology
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Kim KJ, Victor D, Stein E, Valeshabad AK, Saxena P, Singh VK, Lennon AM, Clarke JO, Khashab MA. A novel ballooned-tip percutaneous endoscopic gastrojejunostomy tube: a pilot study. Gastrointest Endosc. 2013 Jul;78(1):154-7. doi: 10.1016/j.gie.2013.03.005. Epub 2013 Apr 24. PMID 23622977

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between 7/1/13 and 4/14/14 in an academic tertiary center
Period: Overall Study
Arm/Group | Self-propelled PEGJ Feeding Tube | Standard PEGJ Feeding Tube
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-propelled PEGJ Feeding Tube | Standard PEGJ Feeding Tube | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.22 (13.30) | 52 (10.68) | 56.84 (12.77)
Sex/Gender, Customized [Number; unit: participants]
  Female | 4 | 8 | 12
  Male | 5 | 2 | 7
Gastrointestinal Quality of Life Index (GIQLI) score [Mean (Standard Deviation); unit: units on a scale] — Gastrointestinal Quality of Life Index (GIQLI) score ranging from 0 (worst quality of life possible with severe digestive symptoms) to 144 (optimal quality of life without symptoms
  units on a scale | 78.2 (27.1) | 69.1 (11.9) | 73.4 (20.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With PEG-J Tube Migration
Description: Number of participants in whom migration was assessed by X-ray at 4 weeks post-intervention.
Time Frame: From date of placement up to 4 weeks
Measure: Number; unit: participants
Arm/Group | Self-propelled PEGJ Feeding Tube | Standard PEGJ Feeding Tube
Number analyzed (Participants) | 9 | 10
participants | 3 | 3

2. Secondary Outcome: Repeat Endoscopy for Feeding Tube Placement Due to Retrograde Tube Migration
Description: Patiens who will have retrograde PEG-J tube migration will get repeat endoscopy for PEG-J tube placement
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Self-propelled PEGJ Feeding Tube | Standard PEGJ Feeding Tube
Number analyzed (Participants) | 9 | 10
participants | 3 | 3

3. Secondary Outcome: Patency of Feeding Tube
Description: Determine tube patency which is defined as time period between tube placement and need for re-intervention.
Time Frame: 2 years
Population: Study terminated prematurely, so that the appropriate follow-up data was not collected.
Arm/Group | Self-propelled PEGJ Feeding Tube | Standard PEGJ Feeding Tube
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Technical Success
Description: Success of tube placement in the desired location as determined endoscopically.
Time Frame: Intra-procedural
Measure: Number; unit: procedure
Arm/Group | Self-propelled PEGJ Feeding Tube | Standard PEGJ Feeding Tube
Number analyzed (Participants) | 9 | 10
procedure | 8 | 10

5. Secondary Outcome: Intervention Time
Description: Time required from introduction of the upper endoscope until placement of the feeding tube.
Time Frame: Intra-procedural
Measure: Mean (Standard Deviation); unit: minute
Arm/Group | Self-propelled PEGJ Feeding Tube | Standard PEGJ Feeding Tube
Number analyzed (Participants) | 9 | 10
minute | 17.2 (12.3) | 28.7 (13.6)

6. Secondary Outcome: Time to Repeat Endoscopy for Tube Replacement
Description: If repeate endocopy and tube placement are needed due to clogging or retrograde migration
Time Frame: 2 years
Population: Study terminated prematurely, so that the appropriate follow-up data was not collected.
Arm/Group | Self-propelled PEGJ Feeding Tube | Standard PEGJ Feeding Tube
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Difficulty of the Procedure
Description: Scored by the endoscopist on a 10-point Visual Analogue Scale with zero being "without difficulty" and 10 being "maximum difficulty".
  The lower the score, the better the outcome.
Time Frame: Inra-procedural
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-propelled PEGJ Feeding Tube | Standard PEGJ Feeding Tube
Number analyzed (Participants) | 9 | 10
units on a scale | 6.2 (3.8) | 7 (2.2)

8. Secondary Outcome: Gastrointestinal Quality of Life Index (GIQLI) Score
Description: Gastrointestinal Quality of Life Index (GIQLI) score ranging from 0 (worst quality of life possible with severe digestive symptoms) to 144 (optimal quality of life without symptoms
Time Frame: 3 month
Population: The discrepancy between the number of analyzed patients and the number of patients in the Participant Flow section is due to the fact that only 5 patients had a completed GIQLI questionnaire at 3-month follow-up.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Self-propelled PEGJ Feeding Tube | Standard PEGJ Feeding Tube
Number analyzed (Participants) | 2 | 3
units on a scale | 106 [72 to 140] | 75 [59 to 80]

9. Secondary Outcome: Short-term Complications
Description: Short-term complications will include stomal (Infection, erythema, bleeding, pain and secretion, etc) and tube (Clotting, dislocation, defect, aspiration, etc) complications detected in the first week.
Time Frame: One week
Measure: Number; unit: participants
Arm/Group | Self-propelled PEGJ Feeding Tube | Standard PEGJ Feeding Tube
Number analyzed (Participants) | 9 | 10
participants | 2 | 3

10. Secondary Outcome: Long-term Complications
Description: Long-term complications will include stomal (Infection, erythema, bleeding, pain, secretion, abscess, etc) and tube (Clotting, dislocation, defect and aspiration, etc) complications detected more than one week after intervention.
Time Frame: 2 years
Population: Study terminated prematurely, so that the appropriate follow-up data was not collected.
Arm/Group | Self-propelled PEGJ Feeding Tube | Standard PEGJ Feeding Tube
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Direct Cost
Description: Cost will be determined according to Medicare reimbursement of billed CPT codes. The cost of all related follow-up procedures will be included (e.g. cost of standard PEGJ in case of failed Self-propelled PEGJ feeding tube, cost of managing complications, cost of re-intervention in case of tube dysfunction, etc)
Time Frame: 2 years
Population: Study terminated prematurely, so that the appropriate follow-up data was not collected.
Arm/Group | Self-propelled PEGJ Feeding Tube | Standard PEGJ Feeding Tube
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Self-propelled PEGJ Feeding Tube | Standard PEGJ Feeding Tube
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 5/9 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Self-propelled PEGJ Feeding Tube (N=9) | Standard PEGJ Feeding Tube (N=10)
Nausea after tube placement (Gastrointestinal disorders) | 5 | 3
vomiting after tube placement (Gastrointestinal disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes